CLINICAL TRIAL: NCT07261410
Title: Active Virtual Reality Distraction on Procedure-Related Emotional Behaviour, Pain, And Anxiety During Venipuncture
Brief Title: Active Virtual Reality Distraction on Procedure-Related Emotional Behaviour, Pain, And Anxiety
Acronym: Oculus2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Proffesor, Pediatric Nursing Department, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VRdeuOculus2
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pain; Anxiety State; Venipuncture
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Standart care
- Active VR (Experimental): The remote control of the virtual glasses will be given to the hand that will not be interfered with, and the child will start, slow down or stop the application herself. Samsung Gear Oculus Guest 2 headset allows watching virtual reality applications.
  Interventions: Device: active VR distraction
- Passive VR (Experimental): It was said that he could watch videos by wearing virtual headset glasses during the procedure. A virtual reality application with Oculus Guest 2 that will attract the attention of children was determined by the researchers.
  Interventions: Device: passive VR distraction

INTERVENTIONS:
Device: active VR distraction — The remote control of the virtual glasses will be given to the hand, and the child will start, slow down or stop the application herself.
  Arms: Active VR
Device: passive VR distraction — watching the application by wearing virtual glasses with Oculus Guest 2
  Arms: Passive VR

SUMMARY:
This study aimed to evaluate the effect of virtual reality methods on procedure-related emotional behaviour, pain, and anxiety levels in school-age children undergoing venipuncture.

DETAILED DESCRIPTION:
Participants were assigned to three groups through stratified randomization: the active VR, the passive VR, and the control group. Children in the VR groups wore VR goggles (Oculus Quest 2) during venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* The child agrees to participate in the study voluntarily.
* The parent agrees to participate in the study voluntarily.
* Obtaining consent forms from the child and parent

Exclusion Criteria:

* The child has a physical and psychological deficit that will prevent him from wearing the glasses that will be placed on his head to watch virtual reality.
* Having fever (>37.5C) and severe dehydration
* The patient did not take analgesics before the intervention

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
procedure related pain | 3 minutes after the phlebotomy
  Wong-Baker FACES (WBS) Pain Rating Scale. This scale uses in children aged 3 and older to rate pain severity, ranges from 0 (very happy/no pain) to 10 (hurts worst).
procedure related anxiety | 3 minutes after the phlebotomy
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
procedure related emotional apperance | immediately after the phlebotomy
  This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'. Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5. The total score is made so that the numerical value is between 5-25 by adding the points obtained for each category. Higher scale score indicates the appearance of more negative emotional behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Prof., Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No